CLINICAL TRIAL: NCT01803529
Title: Standard Heat-pack With or Without Deep Friction Massage for Intercostal Pain in Patients With Heart Disease
Brief Title: Deep Friction Massage for Intercostal Pain in Patients With Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 066-03
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Heart Diseases; Pain
Keywords: thorax; Intercostal Muscles; massage; heat-pack; hot temperature
MeSH Terms: conditions — Heart Diseases; Pain | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- heat-pack with massage (Experimental): deep friction massage and standard heat-pack given a maximum of 8 treatments
  Interventions: Other: heat-pack with massage
- heatpack only (Active Comparator): standard heat-pack given a maximum of 8 treatments
  Interventions: Other: heat-pack only

INTERVENTIONS:
Other: heat-pack with massage
  Arms: heat-pack with massage
Other: heat-pack only
  Arms: heatpack only

SUMMARY:
Studies show that chest pain is a common complaint presented in both general practice and in emergency units. Musculoskeletal causes are common, but frequently overlooked. No studies about treatment of chest pain from the intercostal muscles were found by search in medical literature databases. The purpose of this study is to evaluate the effect of two different physical therapy interventions on intercostal pain in patients with stable heart disease.

The hypothesis was that deep friction massage combined with heat-pack is more effective than heat-pack only.

ELIGIBILITY:
Inclusion Criteria:

* increasing chest pain during a cardiac rehabilitation class
* stable coronary disease
* new re-vascularisation is not planned

Exclusion Criteria:

* unstable coronary disease
* not able to perform the study
* abuse of drugs or alcohol
* participating in other ongoing study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2003-10; Primary Completion 2008-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
pain | 3 months
  Analogue Scale (VAS) 0 to 100, where 0 is no pain and 100 intolerable pains

SECONDARY OUTCOMES:
quality of life | 3 months
  Health-related Quality of life ( HRQL) was evaluated by the disease-specific instrument MacNew and the generic instrument SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Stig A Slørdahl, md prof, Study Director — St. Olavs University Hospital
Locations (1):
- St Olavs University Hospital, Trondheim, Norway

REFERENCES:
- [Result] Berg AT, Stafne SN, Hiller A, Slordahl SA, Aamot IL. Physical therapy intervention in patients with non-cardiac chest pain following a recent cardiac event: A randomized controlled trial. SAGE Open Med. 2015 Apr 16;3:2050312115580799. doi: 10.1177/2050312115580799. eCollection 2015. PMID 26770781